CLINICAL TRIAL: NCT01984255
Title: A Two-Arm, Single Center Pase 1b Trial of Bavituximab Plus Ipilimumab in Advanced Melanoma Patients
Brief Title: A Two-arm, Single Center Phase 1b Trial of Bavituximab Plus Ipilimumab in Advanced Melanoma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: standard of care improved combination treatment of ipilimumab plus nivolumab.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 102013-007; SCCC-05613 (Other: Simmons Cancer Center)
Record Dates: First submitted 2013-10-29; First posted 2013-11-14 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A- Bavituximab plus Ipilimumab (Active Comparator): Arm A-Interventions Drug: Bavituximab Dose:3mg/kg IV over 90 minutes weekly x 2 followed by Bavituximab 3mg/kg IV over 90 minutes weekly Duration-x 12 weeks plus Drug :Ipilimumab 3mg/kg IV over 90 minutes every 3 weeks Duration-x 4.weeks
  Interventions: Drug: Arm A-Bavituximab 3mg/kg IV over 90 minutes weekly x 3 followed by Bavituximab 3mg/kg IV over 90 minutes weekly x 12 plus ipilimumab 3mg/kg IV
- Arm B Ipilimumab (Experimental): Arm B-Interventions Drug- I3mg/kg IV over 90 minutes day 1 followed three weeks later by Drug: Ipilimumab every 3 weeks x 3weeks. Total number of treated patients will be 8.
  Interventions: Drug: Arm B-Ipilimumab 3mg/kg IV over 90 minutes day 1 followed three weeks later by ipilimumab every 3 weeks x 3.

INTERVENTIONS:
Drug: Arm A-Bavituximab 3mg/kg IV over 90 minutes weekly x 3 followed by Bavituximab 3mg/kg IV over 90 minutes weekly x 12 plus ipilimumab 3mg/kg IV — Bavituximab 3mg/kg IV over 90 minutes weekly x 3 followed by Bavituximab 3mg/kg IV over 90 minutes weekly x 12 plus ipilimumab 3mg/kg IV over 90 minutes every 3 weeks x 4. Total number of treated patients will be 16.
  Arms: A- Bavituximab plus Ipilimumab
Drug: Arm B-Ipilimumab 3mg/kg IV over 90 minutes day 1 followed three weeks later by ipilimumab every 3 weeks x 3. — Ipilimumab 3mg/kg IV over 90 minutes day 1 followed three weeks later by ipilimumab every 3 weeks x 3. Total number of treated patients will be 8.
  Arms: Arm B Ipilimumab

SUMMARY:
This is a Open label, two-arm, randomized, two agent, single center trial.

DETAILED DESCRIPTION:
This is a Open label, two-arm, randomized, two agent, single center trial.

Study Product(s), Dose, Route, Regimen:

Bavituximab 3mg/kg IVqwk (IV every week) x 14 plus ipilimumab 3mg/kg IVq3wk (IV every 3 weeks) x 4 or ipilimumab 3mg/kg IVq3wk x 4

Administration Schedule:

Patients will be randomized to one of the following arms:

Arm A-Bavituximab 3mg/kg IV over 90 minutes weekly x 2 followed by Bavituximab 3mg/kg IV over 90 minutes weekly x 12 plus ipilimumab 3mg/kg IV over 90 minutes every 3 weeks x 4. Total number of treated patients will be 16.

Arm B-Arm B-Ipilimumab 3mg/kg IV over 90 minutes day 1 followed three weeks later by ipilimumab every 3 weeks x 3. Total number of treated patients will be 8.

Randomization:

There will be a 2:1 randomization of patients to have a 3 week lead-in treatment with bavituximab followed by combination therapy of ipilimumab + bavituximab versus ipilimumab alone. The assigned treatment will be given once subject is registered successfully.

Endpoints:

Toxicities will be assessed via NCI's CTCAE (Common Terminology Criteria for Adverse Events) v4.1 toxicity criteria. Dose limiting toxicities (DLTs) will be defined as drug-related grade 3-5 adverse events experienced within the first 12 weeks of study treatment. The maximal tolerated dose (MTD) will be exceeded if more than 30% of patients on the study experience DLTs.

DCR will be measured by irRC (Immune-related Complete Response) at weeks 15, 21, 27 using the published algorithm. Disease control rate (DCR) includes complete response (CR), Partial response (PR) and stable disease (SD). Months of survival (MOS) is measured from date of entry into protocol.

Tumor MDSC (Myeloid-Derived Suppressor Cells), TAM and Treg content will be measured by IHC (ImmunoHistoChemistry). Circulating MDSC, TAM and Treg content will be measured by flow cytometry.

Peripheral blood cytokines will be measured by EIA (EIA test is a series of blood tests for diagnosing HIV infection).

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of unresectable or metastatic melanoma. For unknown primary disease, diagnosis of metastatic disease by cytology FNA (Fine Needle Aspiration) is not acceptable.
2. Any number of prior systemic therapeutic regimens including chemotherapy, pathway inhibitors, biochemotherapy, investigational agents, and immunotherapies other than ipilimumab or bavituximab.
3. Subjects must have measurable disease as defined by irRC. All sites must be evaluated within 4 weeks prior to beginning therapy.
4. Age ≥ 18 years.
5. Performance status ECOG (Eastern Cooperative Oncology Group) 0-2.
6. Adequate organ and marrow function as defined below:

   * leukocytes ≥ 2,000/mcL (Microliter)
   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 100,000/mcl
   * total bilirubin < 3X (times) institutional upper limit of normal
   * AST (Aspartate Aminotransferase) (SGOT)/ALT (Alanine Aminotransferase)(SPGT) ≤ 2.5 X institutional upper limit of normal
   * creatinine < 3X institutional upper limit of normal
   * hemoglobin >8g/dL
7. Ability to understand and the willingness to sign a written informed consent.
8. Subjects must be willing to undergo tumor biopsy pretreatment and at weeks 3 and 15.
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

1. No concomitant therapy with any of the following: IL2 (Interleukin 2), interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids; all such therapies must have been discontinued >4weeks.
2. No infection with HIV and no active infection with hepatitis B and no active or chronic infection with hepatitis C. Due to the mechanism of action of ipilimumab, activity and side effects in an immune compromised patient are unknown.
3. Subjects with active CNS (Central nervous system) disease are excluded. Patient with brain metastases previously treated with surgery or stereotactic radiosurgery and with confirmed SD for >8 weeks are allowed.
4. Subjects are excluded if they have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Subjects must not be pregnant or nursing.
7. Any concurrent medical condition requiring the use of systemic steroids is not permitted (the use of inhaled or topic steroids is permitted).
8. Subjects are excluded for receiving any non-oncology vaccine therapy used for prevention of infectious diseases for up to 4 weeks (28 days) prior to or after any dose of ipilimumab.
9. Subjects are excluded if they have a history of prior treatment with ipilimumab, CD137 agonist , CTLA-4 inhibitor (Cytotoxic T-Lymphocyte Antigen 4) or agonist or bavituximab.
10. Patients are excluded if they have a history of autoimmune disease except controlled and stable autoimmune thyroiditis. The excluded autoimmune diseases include acute disseminated encephalomyelitis, Addison's disease, alopecia universalis, ankylosing spondylitis, antiphospholipid antibody syndrome, aplastic anemia, asthma, autoimmune hemolytic anemia, autoimmune hepatitis, autoimmune hypoparathyroidism, autoimmune hypophysitis, autoimmune myocarditis, autoimmune oophoritis, autoimmune orchitis, autoimmune thrombocytopenic purpura, Behcet's disease, bullous pemphigoid, celiac disease, chronic fatigue syndrome, chronic inflammatory demyelinating polyneuropathy, Churg-Strauss syndrome, Crohn's disease, dermatomyositis, dysautonomia, eczema, epidermolysis bullossa acquisita, gestational pemphigoid, giant cell arteritis, Goodpasture's syndrome, Graves' disease, Guillain-Barre syndrome, Hashimoto's disease-except as noted above, IgA nephropathy (Berger's disease), inflammatory bowel disease, interstitial cystitis, Kawasaki's disease, Lambert-Eaton myasthenia syndrome, lupus erythematosis, chronic Lyme disease, Meniere's syndrome, Mooren's ulcer, Morphea, multiple sclerosis, myasthenia gravis, neuromyotonia, opsoclonus myoclonus syndrome, optic neuritis, Ord's thyroiditis, pemphigus, pernicious anemia, polyarteritis nodosa, polyarthritis, polyglandular autoimmune syndrome, primary biliary cirrhosis, psoriasis, Reiter's syndrome, rheumatoid arthritis, sarcoidosis, Sjogren's syndrome, Stiff-Person syndrome, Takayasu's arteritis, ulcerative colitis, Vogt- Kovanagi-Harada disease, vulvodynia, and Wegener's granulomatosis.
11. Subjects are excluded with history of thromboembolic events, clinically significant bleeding-gross hematuria, hemoptysis, or gastrointestinal bleeding, history of bleeding diathesis or hypercoagulable state, ongoing therapy with anticoagulants or non-steroidal anti-inflammatory drugs, or prior exposure to chimeric antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Toxicities | 12 weeks
  Toxicities will be assessed via NCI's CTCAE v4.1 toxicity criteria. Dose limiting toxicities (DLTs) will be defined as drug-related grade 3-5 adverse events experienced within the first 12 weeks of study treatment. The maximal tolerated dose (MTD) will be exceeded if more than 30% of patients on the study experience DLTs.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Months of Survival (measured at weeks 15, 21, and 27)
  DCR will be measured by irRC at weeks 15, 21, 27 using the published algorithm. Disease control rate (DCR) includes complete response (CR), Partial response (PR) and stable disease (SD). Months of survival (MOS) is measured from date of entry into protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Frankel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No